CLINICAL TRIAL: NCT03517085
Title: A Phase 1/2, Open-Label Safety and Dose-Finding Study of Adeno-Associated Virus (AAV) Serotype 8 (AAV8)-Mediated Gene Transfer of Glucose-6- Phosphatase (G6Pase) in Adults With Glycogen Storage Disease Type Ia (GSDIa)
Brief Title: Safety and Dose-Finding Study of DTX401 (AAV8G6PC) in Adults With Glycogen Storage Disease Type Ia (GSDIa)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 401GSDIA01; 1706-1617 (Other: NIH Protocol Registration Number); 2016-003023-30 (EudraCT Number)
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: GSD1
Keywords: glycogen storage disorder Ia; AAV; gene therapy; von Gierke disease; glucose metabolism disorder
MeSH Terms: conditions — Glycogen Storage Disease Type I; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DTX401 Cohort 1 (Experimental): Dose 1 (2.0 × 10^12 GC/kg) with a reactive steroid regimen (6 weeks, at a starting dose of 40 mg/day, after alanine aminotransferase [ALT] elevation)
  Interventions: Genetic: DTX401; Drug: steroid regimen
- DTX401 Cohort 2 (Experimental): Dose 2 (6.0 × 10^12 GC/kg) with a reactive steroid regimen (6 weeks, at a starting dose of 40 mg/day, after ALT elevation)
  Interventions: Genetic: DTX401; Drug: steroid regimen
- DTX401 Cohort 3 (Experimental): Dose 2 (6.0 × 10^12 GC/kg) with an optimized reactive steroid regimen (7 weeks, at a starting dose of 60 mg/day, after ALT elevation)
  Interventions: Genetic: DTX401; Drug: steroid regimen
- DTX401 Cohort 4 (Experimental): Dose 2 (6.0 × 10^12 GC/kg) with a prophylactic steroid regimen (8 weeks, at a starting dose of 60 mg/day, starting on Day 1)
  Interventions: Genetic: DTX401; Drug: steroid regimen

INTERVENTIONS:
Genetic: DTX401 — DTX401 administered as a single peripheral intravenous (IV) infusion
  Other Names: AAV8G6PC; Pariglasgene brecaparvovec
Drug: steroid regimen — prednisone or prednisolone to manage alanine aminotransferase (ALT) elevation

SUMMARY:
The primary objective of the study is to determine the safety of single doses of DTX401, including the incidence of dose-limiting toxicities (DLTs) at each dose level.

DETAILED DESCRIPTION:
Participants enrolled in the 401GSDIA01 study will be monitored for 52 weeks following DTX401 administration. Participants in Cohorts 1, 2, and 3 will receive reactive oral steroid treatment for possible vector-induced hepatitis following treatment with DTX401. Participants in Cohort 4 will receive prophylactic oral steroid treatment to prevent possible vector-induced hepatitis. After completion of the Week 52 visit or early withdrawal, participants will be offered enrollment into a 4-year extension study.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females ≥18 years of age
* Documented GSDIa with confirmation by molecular testing
* Documented history of ≥1 hypoglycemic event with blood glucose <60 mg/dL (<3.33 mmol/L)
* Patient's GSDIa disease is stable as evidenced by no hospitalization for severe hypoglycemia during the 4-week period preceding the screening visit

Key Exclusion Criteria:

* Anti-AAV8 neutralizing antibody titer ≥1:5
* Screening or Baseline (Day 0) blood glucose level <60 mg/dL (<3.33 mmol/L)
* Liver transplant, including hepatocyte cell therapy/transplant
* Presence of liver adenoma >5 cm in size
* Presence of liver adenoma >3 cm and ≤5 cm in size that has a documented annual growth rate of ≥0.5 cm per year
* Significant hepatic inflammation or cirrhosis as evidenced by imaging or any of the following laboratory abnormalities: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN), total bilirubin > 1.5 x ULN, or alkaline phosphatase > 2.5 x ULN

Note additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (6):
- United States (3):
  - UCONN Health, Farmington, Connecticut
  - Michigan Medicine University of Michigan, Ann Arbor, Michigan
  - UT Health - McGovern Medical School, Houston, Texas
- Montreal Children Hospital, McGill University Health Centre, Montreal, Quebec, Canada
- University Medical Center Groningen, Groningen, Netherlands
- Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna, Spain

REFERENCES:
- [Derived] Weinstein DA, Derks TG, Rodriguez-Buritica DF, Ahmad A, Couce ML, Mitchell JJ, Riba-Wolman R, Mount M, Sallago JB, Ross KM, van der Klauw MM, de Boer F, van der Schaaf C, Saavedra H, Martinez-Olmos M, Atanga E, Hosseini A, Mitragotri D, Crombez E. Safety and Efficacy of DTX401, an AAV8-Mediated Liver-Directed Gene Therapy, in Adults With Glycogen Storage Disease Type I a (GSDIa). J Inherit Metab Dis. 2025 Mar;48(2):e70014. doi: 10.1002/jimd.70014. PMID 40064185
- [Derived] Zhang L, Lee C, Arnaoutova I, Anduaga J, Starost MF, Mansfield BC, Chou JY. Gene therapy using a novel G6PC-S298C variant enhances the long-term efficacy for treating glycogen storage disease type Ia. Biochem Biophys Res Commun. 2020 Jun 30;527(3):824-830. doi: 10.1016/j.bbrc.2020.04.124. Epub 2020 May 16. PMID 32430177
- [Derived] Zhang L, Cho JH, Arnaoutova I, Mansfield BC, Chou JY. An evolutionary approach to optimizing glucose-6-phosphatase-alpha enzymatic activity for gene therapy of glycogen storage disease type Ia. J Inherit Metab Dis. 2019 May;42(3):470-479. doi: 10.1002/jimd.12069. Epub 2019 Feb 22. PMID 30714174

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were enrolled sequentially into 4 cohorts of 3 participants each and received a single intravenous (IV) infusion of DTX401, with steroids (prednisone/prednisolone) to manage alanine aminotransferase (ALT) elevation.
Groups:
- DTX401 Cohort 1: DTX401 Dose 1 (2.0 × 10^12 GC/kg) with a reactive steroid regimen (6 weeks, at a starting dose of 40 mg/day, after ALT elevation)
- DTX401 Cohort 2: DTX401 Dose 2 (6.0 × 10^12 GC/kg) with a reactive steroid regimen (6 weeks, at a starting dose of 40 mg/day, after ALT elevation)
- DTX401 Cohort 3: DTX401 Dose 2 (6.0 × 10^12 GC/kg) with an optimized reactive steroid regimen (7 weeks, at a starting dose of 60 mg/day, after ALT elevation)
- DTX401 Cohort 4: DTX401 Dose 2 (6.0 × 10^12 GC/kg) with a prophylactic steroid regimen (8 weeks, at a starting dose of 60 mg/day, starting on Day 1)
Period: Overall Study
Arm/Group | DTX401 Cohort 1 | DTX401 Cohort 2 | DTX401 Cohort 3 | DTX401 Cohort 4
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTX401 Cohort 1 | DTX401 Cohort 2 | DTX401 Cohort 3 | DTX401 Cohort 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (15.3) | 29.7 (10.1) | 26.0 (13.9) | 25.0 (5.2) | 31.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 1 | 4
  Male | 2 | 3 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 3 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Controlled Fasting Challenge: Time to First Hypoglycemic Event [Mean (Standard Deviation); unit: hours] — Time (in hours) to first hypoglycemic event (defined as glucose < 54 mg/dL [< 3.0 mmol/L]) during a controlled fasting challenge.
  hours | 4.4 (0.9) | 4.5 (1.4) | 2.3 (1.2) | 2.5 (0.9) | 3.4 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Treatment-Emergent AEs (TEAEs) Serious TEAEs, Discontinuations Due to TEAEs, and Dose-Limiting Toxicities (DLTs)
Description: An AE is defined as any untoward medical occurrence, regardless of its causal relationship to study product. An SAE is defined as any event that: results in death; is immediately life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; or an important medical event, in the opinion of the investigator. The relationship to study drug was categorized as unrelated, possible, probable or definite. A DLT is defined as any AE/SAE ≥ Grade 3 that is considered by the Investigator and/or Sponsor to be related to DTX401, based on the Nation Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 or later version. Per protocol, SAEs that occurred > 30 days after EOS or Early withdrawal visit, did not need to be reported unless Investigator considered them related to study product.
Time Frame: AEs Prior to Dosing: From signing the informed consent form (ICF) to first dose of study drug. TEAEs: From first dose of study drug through the End of Study (EOS)/Early Withdrawal visit (up to Week 52) plus 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | DTX401 Cohort 1 | DTX401 Cohort 2 | DTX401 Cohort 3 | DTX401 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  Any AE prior to dosing | 1 | 1 | 2 | 2
  Any TEAE | 3 | 3 | 3 | 3
  Related TEAE | 3 | 3 | 3 | 3
  Serious TEAE | 2 | 1 | 1 | 0
  Serious related TEAE | 0 | 0 | 0 | 0
  Grade 3 or 4 TEAE | 0 | 0 | 1 | 0
  Dose-limiting toxicity | 0 | 0 | 0 | 0
  TEAE leading to study discontinuation | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Time to First Hypoglycemic Event Over Time
Description: The change from baseline in time (in hours) to first hypoglycemic event (defined as glucose < 54 mg/dL [< 3.0 mmol/L]) during a controlled fasting challenge at 12, 24, and 52 weeks after IV administration of DTX401. A positive change from baseline is favorable.
Time Frame: Baseline, Weeks 12, 24, 52
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DTX401 Cohort 1 | DTX401 Cohort 2 | DTX401 Cohort 3 | DTX401 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
hours
  Change at Week 12: number analyzed (Participants) | 3 | 3 | 3 | 0
  Change at Week 12 | 3.3 (2.0) | 1.7 (0.6) | 1.4 (0.8) |
  Change at Week 24: number analyzed (Participants) | 3 | 3 | 3 | 1
  Change at Week 24 | 4.3 (4.2) | 0.5 (0.6) | 0.7 (1.7) | 0.3 (NA) — 1 participant analyzed
  Change at Week 52: number analyzed (Participants) | 3 | 3 | 2 | 3
  Change at Week 52 | 4.2 (2.2) | -1.8 (1.7) | -0.6 (0.1) | 3.6 (2.7)

ADVERSE EVENTS:
Time Frame: From enrollment (all-cause mortality) or first dose of study drug (treatment emergent adverse events) through the End of Study/Early Withdrawal visit (up to Week 52) plus 30 days.
Description: Per protocol, SAEs that occurred > 30 days after EOS or Early withdrawal visit, did not need to be reported unless Investigator considered them related to study product.
Groups:
- Total: DTX401 Dose 1 (2.0 × 10^12 GC/kg) or DTX401 Dose 2 (6.0 × 10^12 GC/kg) with a reactive steroid regimen (6 weeks, at a starting dose of 40 mg/day, after ALT elevation), an optimized reactive steroid regimen (7 weeks, at a starting dose of 60 mg/day, after ALT elevation), or a prophylactic steroid regimen (8 weeks, at a starting dose of 60 mg/day, starting on Day 1)
Arm/Group | DTX401 Cohort 1 | DTX401 Cohort 2 | DTX401 Cohort 3 | DTX401 Cohort 4 | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 0/3 | 4/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTX401 Cohort 1 (N=3) | DTX401 Cohort 2 (N=3) | DTX401 Cohort 3 (N=3) | DTX401 Cohort 4 (N=3) | Total (N=12)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Metabolic Disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTX401 Cohort 1 (N=3) | DTX401 Cohort 2 (N=3) | DTX401 Cohort 3 (N=3) | DTX401 Cohort 4 (N=3) | Total (N=12)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 1
Adrenal Suppression (Endocrine disorders) | 0 | 0 | 1 | 0 | 1
Glucocorticoid Deficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 0 | 0 | 1
Face Oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 2
Hunger (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Thirst (General disorders) | 1 | 0 | 0 | 0 | 1
Hepatic Pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Food Allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0 | 2
Abdominal Wall Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sinobronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Tinea Pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1 | 0 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Stoma Site Discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 2 | 2 | 2 | 6
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 0 | 2
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 2 | 1 | 0 | 4
Blood Creatinine Increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood Glucose Fluctuation (Investigations) | 0 | 0 | 2 | 0 | 2
Blood Uric Acid Increased (Investigations) | 0 | 0 | 1 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 1 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 1 | 0 | 2
Liver Function Test Increased (Investigations) | 2 | 1 | 0 | 0 | 3
Weight Decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 4
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Joint Noise (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 2 | 1 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Libido Increased (Psychiatric disorders) | 2 | 0 | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 2
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 3
Skin Striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03517085/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT03517085/SAP_001.pdf